CLINICAL TRIAL: NCT03242135
Title: Role of Red Cell Distribution Width as Anon Invasive Index for Predicting Liver Cell Failure and Portal Hypertension in Cirrhotic Patient
Brief Title: Role of RDW as Anon Invasive Index for Predicting Liver Cell Failure and Portal Hypertension in Cirrhotic Patient
Acronym: RDW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Atef, Principal Investigator, Assiut University
Other Study IDs: 17100264
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Predicting Liver Cell Failure & Portal Hypertension in LC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
role of RDW as anon invasive method for predicting liver cell failure & portal hypertension in cirrhotic patient

DETAILED DESCRIPTION:
Red blood cell distribution width (RDW) is a measure of the range of variation of red blood cell (RBC) volume. The RDW-SD (Standard deviation ) is an actual measure of size. Normal reference range of RDW-SD in adult human is 39-46 fL .Liver plays an important role in removing body toxins which affects RBCs ,so liver cirrhosis may affects the RDW. Cirrhosis is a chronic degenerative disease in which irreversible scarring of the liver occurs. It leads to liver failure. Child's score is used as an indicator for liver cell function Portal hypertension is an increase in the blood pressure within the portal venous system .Obstruction to blood flow that occurs in liver due to fibrosis and regenerating nodules reduce flow from the portal veins into the hepatic veins. It also impedes hepatic artery flow from the branches that feed into the sinusoids. This increase in arterial resistance leads to an increase in arterial flow into the portal vein via producing a new anastamosis. The net result of that is an increase in portal vein pressure and dilatation of portal vein. Direct measurement of portal pressure is invasive, inconvenient, and clinically impractical. The Hepatic Venous Pressure Gradient (HVPG) is used to measure portal pressure .Recently, portal vein diameter is used as indicator for portal hypertension .

ELIGIBILITY:
Inclusion Criteria:

The study will include a total of 100 patient in Assiut university hospital diagnosed to be cirrhotic by abdominal US. They will be divided into 3 groups according to Child's score (A,B,C)

Exclusion Criteria:

* Evidence of iron deficiency anaemia
* Patients within one month of hematemesis
* Thalassaemia

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include a total of 100 patient in Assiut university hospital diagnosed to be cirrhotic by abdominal US
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09-21 (Actual); Primary Completion 2018-02-21 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Role of RDW (red cell distribution width) as a non invasive index for predicting liver cell failure and portal hypertension in cirrhotic patient | 3 years
  To develop a simple predictive method for liver cell failure and portal hypertension in cirrhotic patient using the routine hematological parameters (RDW in complete blood count ) & abdominal US

CONTACTS AND LOCATIONS:
Overall Officials: marina Atef, master, Principal Investigator — Assiut University
Locations (1):
- Marina Atef, Asyut, Egypt